CLINICAL TRIAL: NCT06316505
Title: Use of Oral Photographs of Patients on Oral Hygiene Motivation Promotes Periodontal Health: a Prospective Randomized Controlled Trial
Brief Title: Oral Photographs of Patients on Oral Hygiene Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Didem OZKAL EMINOGLU (Other)
Responsible Party: Sponsor-Investigator, Didem OZKAL EMINOGLU, assistant professor, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 11/2023-58
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Periodontal Diseases; Motivation; Hygiene
Keywords: oral hygiene; periodontal health; periodontal indices; motivation; Modified Bass Technique
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (CG) (No Intervention): Conventional oral hygiene education (COHE)
- Intervention group (IG) (Experimental): In addition to COHE, oral hygiene motivation with individual oral photographs
  Interventions: Behavioral: Oral hygiene motivation with individual oral photograps

INTERVENTIONS:
Behavioral: Oral hygiene motivation with individual oral photograps — Oral photograps was taken at control sessions.
  Arms: Intervention group (IG)

SUMMARY:
Based on these considerations, this randomized controlled trial aimed to determine the effectiveness of a personalized visual oral health education program in addition to conventional education on oral hygiene by comparing changes in clinical periodontal parameters.

Participants will get conventional oral hygiene education (COHE) with/without visual motivation using self oral photographs of patients.

Researchers will compare Intervention group and control groups on oral hygiene by comparing changes in clinical periodontal parameters.

DETAILED DESCRIPTION:
Maintaining oral health requires a motivated patient. The adherence to a lifelong oral hygiene regimen is significantly influenced by an individual's motivation and manual dexterity. The physician's responsibility in this context is to provide guidance to the patient regarding the appropriate and efficient oral hygiene routine, as well as to motivate their adherence to it. The definition of motivation is to stimulate action or effort towards a particular goal or objective. Motivation is a condition that can be altered in response to external influences and time, rather than being a characteristic. The primary objective of motivation is to enhance persons' knowledge of this matter by highlighting oral health, introducing oral hygiene, and offering information on efficacious mechanical cleaning procedures for eliminating factors that contribute to the deterioration of oral hygiene.

Participants were divided into 2 groups using https://www.randomizer.org/ website:

Control group (CG) (n=28): Conventional oral hygiene education (COHE) [22]

Intervention group (IG) (n=28): In addition to COHE, the following steps were followed:

* Session 1: A photograph was taken before (F1) and after (F2) full-mouth scaling root planing (fmSRP). Then the patient was shown the difference.
* 2nd session: A photograph was taken (F3) and the patient is shown the difference between F1 and F3.
* 3rd session: A photograph was taken (F4) and the patient is shown the difference between F1 - F3 - F4.

ELIGIBILITY:
Inclusion Criteria:

* age ranging from 18-60 years;
* a minimum of 12 teeth;
* and being available for the follow-up assessment
* participants were wanted to be right-handers when toothbrushing to standardization.

Exclusion Criteria:

* Patients with systemic illnesses or conditions,
* smokers and individuals taking any medication that may affect periodontal health were not included in the study.
* Individuals who had previously been treated for periodontal disease in the past 6 months were also excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Clinical periodontal parameters / plaque index (PI) | T0: baseline, T1: 1 month after baseline, T2: 3 months after baseline
  The amount of plaque present on the teeth was assessed using a plaque staining agent and graded according to the plaque index system. Higher scores mean a worse outcome.
Clinical periodontal parameters / gingival index (GI) | T0: baseline, T1: 1 month after baseline, T2: 3 months after baseline
  The presence and extent of gingival inflammation and bleeding were graded according to the gingival index system. Higher scores mean a worse outcome.
Clinical periodontal parameters / probing pocket depth (PPD). | T0: baseline, T1: 1 month after baseline, T2: 3 months after baseline
  PPD was measured as the distance between the deepest point of the sulcus and the gingival margin. Higher scores mean a worse outcome.
Clinical periodontal parameters / bleeding on probing (BOP) | T0: baseline, T1: 1 month after baseline, T2: 3 months after baseline
  The presence of bleeding on probing is considered an objective sign of periodontal inflammation. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: DİDEM ÖZKAL EMİNOĞLU, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozkal Eminoglu D, Sahin BN, Bicer D, Dal G, Huseynli I, Dadashov A, Betul Dogan D, Kasali K. Using patients' oral photographs for oral hygiene motivation promotes periodontal health: a prospective randomized controlled trial. BMC Oral Health. 2024 Jul 13;24(1):786. doi: 10.1186/s12903-024-04553-7. PMID 38997684